CLINICAL TRIAL: NCT06694935
Title: A Phase 1b Study of QX1206 in Type 2 Diabetes Mellitus (T2DM) Patients With Non-Alcoholic Fatty Liver Disease (NAFLD)
Brief Title: A Phase 1b Study of QX1206 in T2DM Patients With NAFLD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: 1Globe Health Institute (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2DM-QX1206-1
Record Dates: First submitted 2024-11-04; First posted 2024-11-19 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Non-Alcoholic Fatty Liver Disease (NAFLD)
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QX1206 (Experimental)
  Interventions: Drug: QX1206

INTERVENTIONS:
Drug: QX1206 — QX1206 will be administered orally before bedtime

SUMMARY:
This is an open label phase 1b trial of QX1206 in patients with T2DM and with NAFLD. Laboratory tests and other measurements will be assessed prior to the first dose of study treatment and throughout the study to determine the recommended phase 2 dose. In addition, the preliminary effects of QX1206 on antidiabetic activity and other metabolic parameters will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent must be obtained and documented
* 18 years of age and < 65 years old
* BMI ≥ 18 kg/m^2 and < 45 kg/m^2
* T2DM diagnosed per 2021 American Diabetes Association criteria
* Diagnosis of NAFLD
* For male or female patients of child producing potential: must agree to use contraception or take measures to avoid pregnancy during the study
* Women of child-bearing potential (WOCBP) must have a negative pregnancy test
* Serum creatinine < 1.5×ULN or creatinine clearance ≥ 60 ml/min
* Participating patients must be able to comply with all study requirements and the study center must have appropriate means of ensuring protocol compliance for each participating patient

Exclusion Criteria:

* Uncontrolled diabetes
* Patients with an active, serious medical disease that limit activities of daily living
* Patients with current, significant alcohol consumption or a history of significant alcohol consumption
* Patients with any of the following clinical laboratory abnormalities at screen and confirmed by a single repeat if deemed necessary:
* Fasting triglycerides > 500 mg/dL
* Fasting direct LDL-C > 190 mg/dL
* AST > 5.0 × upper limit of normal (ULN)
* ALT > 5.0 × ULN
* Alkaline phosphatase (ALP) ≥ 2 × ULN
* HbA1c > 10.5%
* Fasting plasma glucose (FPG) > 240 mg/dL (13.3 mmol/L)
* Platelets count < 140,000/mm^3
* Patient takes drugs historically associated with NAFLD and other known hepatotoxins
* Treatment with drugs (e.g., vitamin E > 400 IU/day) or herbal supplements with potential anti-NAFLD effect

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | Baseline Day 1 up to Week 12

SECONDARY OUTCOMES:
Hemoglobin A1c (HbA1c) | 12 Weeks
  Change in HbA1c percentage from baseline with QX1206
Fasting plasma glucose (FPG) | 12 Weeks
  Change in FPG mg/dL from baseline with QX1206
Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) | 12 Weeks
  Change in the HOMA-IR from baseline with QX1206
Fasting insulin | 12 Weeks
  Change in fasting insulin pmol/L from baseline with QX1206

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Keates, PhD, Study Director — 1Globe Health Institute
Locations (1):
- Centricity Research Toronto LMC., Toronto, Canada